CLINICAL TRIAL: NCT03426735
Title: Multicenter Study to Evaluate the Effectiveness of Dry Heat in the Extravasations of Iodinated Contrast.
Brief Title: Study of Iodine Contrast Media Extravasation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Sant Pau (Other)
Collaborators: University of Barcelona (Other)
Responsible Party: Principal Investigator, Jaume Roca Sarsanedas, Radiology Nurse, Hospital de Sant Pau
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC/16/258/4709
Record Dates: First submitted 2018-01-29; First posted 2018-02-08 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Contrast Media Extravasation
Keywords: Iodine; Iodized; Computerized Tomography; Extravasation; contrast media
MeSH Terms: conditions — Extravasation of Diagnostic and Therapeutic Materials

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry heat (Experimental): Dry heat application with a termal bag
  Interventions: Other: Dry heat
- Dry cold (Active Comparator): Dry cold application with a termal bag
  Interventions: Other: Dry cold

INTERVENTIONS:
Other: Dry heat — Dry heat will be applied in the extravasation zone for 10 minutes. Let it rest for 20 and proceed to make a second application of dry cold for another 10 minutes. The control is after 24 hours.
  Arms: Dry heat
Other: Dry cold — Dry cold will be applied in the extravasation zone for 10 minutes. Let it rest for 20 and proceed to make a second application of dry cold for another 10 minutes. The control is after 24 hours.
  Arms: Dry cold

SUMMARY:
The purpose of this study is to determine the best intervention after the extravasation of the iodinated contrast medium out of a vessel into the surrounding tissues.

DETAILED DESCRIPTION:
The risk of intravenous extravasation of iodinated contrast media has a relatively low incidence, although the increase in requests for computed tomography scans where it can manage contrasts with a large volume, high osmolality, high-speed injection pumps and even with an added electrical load, has caused an increase in this risk and its complications.

When there is an extravasation of iodinated contrast medium, in most published recommendations and guidelines advise local conservative measures, but there is no consensus on whether cold or heat should be applied as the first intervention to minimize the consequences and favour a rapid resolution.

This study aims to evaluate the effectiveness of the application of heat in the extravasations of iodinated contrast, providing the necessary evidence to determine the best cure that can be applied in the current circumstances of administration, by injection pumps at high speeds and large volumes.

ELIGIBILITY:
Inclusion Criteria:

* Computed tomography procedure.
* Administration of the contrast medium with injection pump between 1,5 and 8 ml/s.
* Peripheral venous access in the arms or legs.

Exclusion Criteria:

* Administration of the contrast medium with central venous access.
* Renal insufficiency.
* Iodine allergy.
* Immediate acute complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Time resolution the swelling and pain. | 24-48 hours past

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - Hospital General de l´Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Health Diagnostic General Catalunya, Sant Cugat del Vallès, Barcelona
  - Hospital de Sant Joan Despí Moisès Broggi, Sant Joan Despí, Barcelona
  - Radiología del Parc Salut Mar, Barcelona
  - Health Diagnostic Teknon, Barcelona
  - Servicio Radiologia Clínica Sagrada Familia, Barcelona
  - Health Diagnostics Sagrat Cor, Barcelona
  - Centre de Diagnòstic per la Imatge Clínic, Barcelona
  - Hospital Sant Pau, Barcelona